CLINICAL TRIAL: NCT00242619
Title: Rosiglitazone Add-On in Treatment of Depressed Patients With Insulin Resistance: a Pilot Study
Brief Title: Insulin Resistance in Patients With Mood Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Natalie Rasgon, Principal Investigator, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 95552
Record Dates: First submitted 2005-10-19; First posted 2005-10-20 (Estimated); Results first posted 2017-02-14 (Actual); Last update posted 2017-02-14 (Actual); Status verified 2016-12

CONDITIONS: Depression; Bipolar Disorder; Insulin Resistance
MeSH Terms: conditions — Depression; Bipolar Disorder; Insulin Resistance | interventions — Rosiglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rosiglitzone (Experimental): This group includes all 12 subjects who received rosiglitazone. Rosiglitazone was administered in addition to current antidepressant and/or mood-stabilizing medication at a dose of 4 mg/day for the first 4 weeks, with subsequent increase in dose to 9 mg/day for the remaining 8 weeks of the 12-week trial.
  Interventions: Drug: rosiglitazone

INTERVENTIONS:
Drug: rosiglitazone — Rosiglitazone was administered at two different doses over the 12-week period.
  Other Names: Avandia

SUMMARY:
Insulin resistance is known to be associated with mood disorders and cognitive difficulties. The purpose of this study is to treat depressed patients with rosiglitazone (also known as [AKA] Avandia), therefore improving glucose sensitivity, which in turn has the potential to affect mood and thinking. We, the researchers at Stanford University, are recruiting men and women who have been diagnosed with depression, and are willing to participate in this 3 month study. Participation involves neuropsychological testing, 2 blood draws called an oral glucose tolerance test (OGTT), which tests for glucose and insulin levels, and the medication, rosiglitazone. Participants are allowed to continue on their current psychiatric medication.

DETAILED DESCRIPTION:
An association between insulin resistance (IR) and affective disorders has been postulated in a number of cross-sectional studies. Limited data exist on potential changes in IR associated with improvement in depressive symptoms and/or depression remission resolution - two studies reported decreased IR after successful antidepressant treatment, while another study reported persisting IR even after successful treatment.

We have postulated that IR is a part of the pathophysiology of affective disorders, and its improvement (via pharmacological or nonpharmacological treatments) may significantly reduce the severity of depressive symptoms. In support of this hypothesis, we previously reported increased IR in women with bipolar disorder, as well as a significant association between IR and depressive symptoms in women with primary IR syndrome (polycystic ovary syndrome [PCOS]). In the current pilot study, we attempted a more direct testing of the hypothesis that improvement of IR will result in improvement in mood in patients with depressive disorders. The aim of the study was to evaluate whether addition of the peroxisome proliferator-activated receptor-γ (PPAR) agonist rosiglitazone to the treatment as usual (TAU) of nondiabetic patients with unipolar or bipolar depression would result in improvement in depression severity and clinical global impression (CGI). Insulin sensitizing agents have proven efficacious in nondiabetic IR, or "prediabetic", individuals. All subjects in this pilot study had elevated fasting plasma glucose (FPG) and ratios of high density lipoproteins (HDL) to triglycerides (TG), which are established surrogate markers of IR.

In the current pilot study, we attempted a more direct testing of the hypothesis that improvement of IR will result in improvement in mood in patients with depressive disorders. The aim of the study was to evaluate whether addition of the peroxisome proliferator-activated receptor-γ (PPAR) agonist rosiglitazone to the treatment as usual (TAU) of nondiabetic patients with unipolar or bipolar depression would result in improvement in depression severity and clinical global impression (CGI). Insulin sensitizing agents have proven efficacious in nondiabetic IR, or "prediabetic", individuals. All subjects in this pilot study had elevated fasting plasma glucose (FPG) and ratios of high density lipoproteins (HDL) to triglycerides (TG), which are established surrogate markers of IR.

ELIGIBILITY:
Inclusion Criteria:- Current depression

* Insulin resistance
* Current physician/psychiatrist care
* Between the ages of 18-60
* Willing to sign the Human Subjects Protection Consent Form
* Willing to have blood sampling Exclusion Criteria:- Diabetes
* History of unstable heat disease
* Uncontrolled hypertension
* Extensive use of alcohol
* Current use of street drugs
* History of myocardial infarction
* History of cerebrovascular disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2007-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Natalie Rasgon, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Completers: Subjects who completed the study and 12 weeks of taking rosiglitazone.
- Drop-Outs: Subjects who dropped out and did not complete the 12 weeks on rosiglitazone.
Period: Overall Study
Arm/Group | Completers | Drop-Outs
Started | 8 | 4
Completed | 8 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Completers: Subjects who met all criteria, took rosiglitazone, and completed the study.
- Drop-Outs: Subjects who met all criteria, took rosiglitazone, and did not complete the study.
- Total: Total of all reporting groups
Arm/Group | Completers | Drop-Outs | Total
Number analyzed (Participants) | 8 | 4 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 4 | 12
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (5.6) | 52.0 (6.5) | 51.95 (6.05)
Gender [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 8 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression Rating Scale (HDRS-21)
Description: The Hamilton Depression Rating Scale (HDRS-21) measures depression severity on a scale from 0 to 21, with 0 being the lowest level of depression severity and 21 being the highest level of depression severity.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Completers: Subjects who completed the study.
- Drop-Outs: Subjects who dropped out of the study.
Arm/Group | Completers | Drop-Outs
Number analyzed (Participants) | 8 | 4
units on a scale | 19.9 (5.0) | 13.0 (0.8)

2. Primary Outcome: Clinical Global Impression-Severity Scale (CGI-S)
Description: The Clinical Global Impression-Severity Scale (CGI-S) assesses depression severity. It is a 7-point scale, where 1 is the lowest level of depression severity and 7 is the highest level of depression severity.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Completers | Drop-Outs
Number analyzed (Participants) | 8 | 4
units on a scale | 4.1 (0.6) | 3.3 (0.5)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over 12 weeks.
Arm/Group | Completers | Drop-Outs
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/4
Other Adverse Events (participants affected / at risk) | 0/8 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No